CLINICAL TRIAL: NCT05460559
Title: Endoscopic Combined Intrarenal Surgery Versus Multi-Tract Percutaneous Nephrolithotomy for Complex Renal Stones: A Randomized Controlled Trial
Brief Title: Endoscopic Combined Intrarenal Surgery Versus Multi-Tract Percutaneous Nephrolithotomy for Complex Renal Stones:
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Abdel-Lateif El-Sawy, Lecturer of Urology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AS-7-2022
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Stone, Kidney
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (p-PCNL) procedure (Active Comparator): In lithotomy position, . Under fluoroscopic guidance, the desired calyces will be punctured using an 18 G coaxial needle. Then 0.038 mm hydrophilic guidewires will be passed percutaneously through the needle into the pelvis. Using metal dilators dilatation will be carried out. Amplatz sheath will be inserted to allow nephroscope to enter the collecting system. Stone disintegration will be performed using pneumatic, ultrasonic or laser lithotripsy. Eventually after removal of all stone fragments, a nephrostomy tube will be placed.
  Interventions: Procedure: Group A (p-PCNL) procedure
- Group B (s-ECIRS) procedure (Experimental): The patients will be in Galdakao-Modified Supine Valdivia (GMSV) position . Under fluoroscopic guidance, the desired calyces will be punctured using an 18 G coaxial needle. Then 0.038 mm hydrophilic guidewires will be passed percutaneously through the needle into the pelvis. Using metal dilators dilatation will be carried out till 30 Fr. Amplatz sheath will be inserted to allow a 26 Fr nephroscope to enter the collecting system. Retrograde intrarenal surgery will be applied simultaneously by a second surgeon using flexible ureteroscopy. The stones will be fragmented with holmium-yttrium-aluminum-garnet (YAG) laser and stone fragments will be evacuated by basket or removed through PCNL tract under nephroscopy.
  Interventions: Procedure: Group B (s-ECIRS) procedure

INTERVENTIONS:
Procedure: Group A (p-PCNL) procedure — In lithotomy position, ureteric catheter will be inserted allowing injection of contrast to obtain a pyelogram. Shifting the patients in prone position will be done. Under fluoroscopic guidance, the desired calyces will be punctured using an 18 G coaxial needle. Then 0.038 mm hydrophilic guidewires will be passed percutaneously through the needle into the pelvis. Using metal dilators dilatation will be carried out. Amplatz sheath will be inserted to allow nephroscope to enter the collecting system. Stone disintegration will be performed using pneumatic, ultrasonic or laser lithotripsy. Eventually after removal of all stone fragments, a nephrostomy tube will be placed.
  Arms: Group A (p-PCNL) procedure
Procedure: Group B (s-ECIRS) procedure — The patients will be in Galdakao-Modified Supine Valdivia (GMSV) position . Under fluoroscopic guidance, the desired calyces will be punctured using an 18 G coaxial needle. Then 0.038 mm hydrophilic guidewires will be passed percutaneously through the needle into the pelvis. Using metal dilators dilatation will be carried out till 30 Fr. Amplatz sheath will be inserted to allow a 26 Fr nephroscope to enter the collecting system. Retrograde intrarenal surgery will be applied simultaneously by a second surgeon using flexible ureteroscopy. The stones will be fragmented with holmium-yttrium-aluminum-garnet (YAG) laser and stone fragments will be evacuated by basket or removed through PCNL tract under nephroscopy.
  Arms: Group B (s-ECIRS) procedure

SUMMARY:
The aim of this study is to compare outcomes of endoscopic combined intrarenal surgery (ECIRS) with the multi-tract percutaneous nephrolithotomy for management of complex renal stones.

DETAILED DESCRIPTION:
Nephrolithiasis is a very common disease and continues to be a common cause of morbidity. The evolving epidemiology of this disease includes changes in gender distribution and associations with systemic disease. The currently available modalities for the treatment of renal calculi include extracorporeal shockwaves lithotripsy (SWL), flexible ureteroscopy (FURS) and percutaneous nephrolithotomy (PCNL).

Complex renal stones usually refer to multiple stones, stones associated with anatomical or functional abnormalities or staghorn calculi. They can cause severe morbidities such as renal failure, sepsis, and even death. Rassweiler et al. defined complex renal calculi based on stone burden and distribution, renal function and associated infection. Due to the complicated etiological factors, large stone burdens, high operation risks and high recurrence, it is always a challenge for surgeons to treat such stones. Complete stone clearance is the ultimate goal in staghorn calculi management because of the high incidence of recurrence and its inherent risks to the kidney and life of the patient.

Various management options are available for management of staghorn renal calculi including PCNL monotherapy, single-tract PCNL with flexible nephroscopy, multi-tract PCNL, combinations of PCNL and SWL, SWL monotherapy and open surgical options.

The American Urological Association (AUA) guidelines recommend PCNL as the first-line treatment for staghorn calculi. According to the European Association of Urology (EAU) guidelines, SWL remains the method of choice for the removal of stones within the renal pelvis, upper or middle calices measuring < 2 cm while larger stones (more than 2 cm) and lower pole stones more than 1.5 cm should be managed using PCNL.

It is noteworthy that prone position is conventionally used for PCNL surgical procedure, which facilitates percutaneous renal puncture and decreases the chance of splanchnic injury. However, it confines the application of Endoscopic Combined Intra-Renal Surgery (ECIRS). Scoffone CM et al. reported the use of ECIRS in Galdakao-Modified Supine Valdivia (GMSV) position for complex urolithiasis, the results showed that ECIRS in GMSV position generated high one step SFR, without additional procedure related complications.

As stone size increases, longer operative time, larger volume of irrigating fluid and multiple tracts may be required to achieve complete stone clearance as it is very difficult to access all the calices through a single percutaneous tract. Multiple access tracts are needed in as many as 20% to 58% of PCNL procedures.In case of complex calculi, the number of accesses is defined by the overall size, volume of the stone, anatomy of the pelvi-calyceal system (PCS), stone distribution, general health of the patient and the experience of the operating surgeon. So, multi-tract PCNL has been well established in the management of complex renal calculi. El-Nahas AR et al. reported that with PCNL monotherapy, the stone free rate (SFR) for staghorn calculi was 56%.Multiple tracts or multiple sessions of PCNL were required to get high SFR in patients with staghorn calculi while the tract related complications increased accordingly such as extravasation, bleeding, need for transfusion, infection, fever and deterioration in renal function. Indeed, several investigators have reported greater blood loss with more than one access tract.

On the other hand, many evidences have demonstrated that FURS is effective and safe for the renal stone less than 2 cm. Recently it is used to treat relatively large size intrarenal calculi . A meta-analysis published in 2012 showed that FURS can successfully treat patients with renal stones > 2 cm with satisfactory clinical outcome. However, flexible ureteroscopic lithotripsy is not recommended as monotherapy for staghorn calculi, while an important ancillary therapeutic option for residual stones following PCNL.

So, we need a new treatment modality to minimize the morbidity of multi-tract PCNL by evaluation of the ECIRS.

ELIGIBILITY:
Inclusion Criteria:

* Patients' age ≥ 18 years.
* Patients who are diagnosed as complex renal calculi (Guy's Stone Score (GSS) 3 or 4) as detected by Non-contrast Computed Tomography (NCCT).

Exclusion Criteria:

* Renal anatomic anomalies.
* Solitary kidney.
* Coagulation disorders.
* Skeletal deformity.
* Active urinary tract infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
One stage stone free rate | first post-operative day
  It will include the one-stage SFR which is defined as the number of patients who will show no residual stones or only residual stone fragments < 4 mm in diameter at postoperative day-1 assessment NCCT

SECONDARY OUTCOMES:
Number of percutaneous access tracts required. | during the procedure
  Number of percutaneous access tracts required.
Postoperative complications | 30 days after intervention
  Postoperative complications (Type, rate and using modified Dindo-Clavian grading system).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A El-Nahas, Study Director — Mansoura University; Ahmed A Elshal, Study Director — Mansoura University
Locations (1):
- Mansoura Urology and Nephrology Center, Al Mansurah, Outside U.S./Canada, Egypt

IPD SHARING:
Plan to Share IPD: No